Trial Title: Oxford Acute Myocardial Infarction - Pressure-controlled Intermittent Coronary Sinus Occlusion in STEMI (OxAMI-PICSO study)

## NCT03473015

Ethics Ref: 15/SC0167

Date and Version No: 26 February 2018 Version 5.0

Chief Investigator: Prof. Adrian Banning (Oxford University Hospital)

**Investigators:** Prof. Keith Channon (University of Oxford)

Dr. Raj Kharbanda (Oxford University Hospitals)

Dr. Colin Forfar (Oxford University Hospitals)

Prof. Stefan Neubauer (University of Oxford)

Prof. Robin Choudhury (University of Oxford)

Dr. Giovanni Luigi De Maria (University of Oxford)

Dr. Erica Dall'Armellina (University of Oxford)

Dr. Vanessa Ferreira (University of Oxford)

**Sponsor:** Oxford University Hospitals NHS Trust

**Funders:** Miracor Medical Systems

BRC ACS theme

## **Chief Investigator Signature:**

## No potential conflicts of interest to declare

# **Confidentiality Statement**

This document contains confidential information that must not be disclosed to anyone other than the Sponsor, the Investigator Team, host organisation, and members of the Research Ethics Committee, unless authorised to do so.

# **TABLE OF CONTENTS**

| 1. | KEY TRIAL CONTACTS | 4 |
|---|---|---|
| 2. | SYNOPSIS | 4 |
| 3. | ABBREVIATIONS | 6 |
| 4. | BACKGROUND AND RATIONALE | 7 |
| 5. | OBJECTIVES AND OUTCOME MEASURES/ENDPOINTS | 11 |
| 6. | TRIAL DESIGN | 12 |
| 7. | PARTICIPANT IDENTIFICATION | 13 |
| 7.1. | Trial Participants | 13 |
| 7.2. | Inclusion Criteria | 14 |
| 7.3. | Exclusion Criteria | 14 |
| 8. | TRIAL PROCEDURES | 15 |
| 8.1. | Informed Consent | 15 |
| 8.2. | Discontinuation/Withdrawal of Participants from Trial Treatment | 19 |
| 8.2.1 | Study Withdrawal | 19 |
| 8.2. | .2 Participant death: | 19 |
| 8.3 | Study timeline (see "Integrated flowchart for OxAMI-PICSO study" as below) | 19 |
| 8.3. | .1 Stage 1: Pre-Stenting | 20 |
| 8.3. | .2 Stage 2: PICSO treatment | 21 |
| 8.3. | .3 Stage 3: Stenting | 21 |
| 8.3. | .4 Stage 4: 24-48 hours post PCI | 22 |
| 8.3. | .5 Stage 5: 6 months post PCI | 22 |
| 8.4 | Definition of End of Trial | 23 |
| 9. | STUDY ASSESSMENT | 23 |
| 9.1 | Data Collection, Patient Reported Outcomes and Cardiovascular Outcomes | 23 |
| 9.2 | PICSO device | 23 |
| 9.3 A | nalysis of CMR | 23 |
| 9.4 A | nalysis of cardiac physiological measurements | 23 |
| 10. | IDENTIFICATION & DESCRIPTION OF THE INVESTIGATIONAL DEVICE | 25 |
| 10.1 | Device description | 25 |
| 10.2 | Device Safety | 27 |
| 10.3 | Device Accountability | 29 |
| 11 | SAFETY REPORTING | 29 |
| 11 1 | Definitions | 29 |

| 11.2 | Causality | 32 |
|---|---|---|
| 11.3 | Procedures for Recording Adverse Events | 33 |
| 11.4 | Reporting Procedures for Serious Adverse Events | 34 |
| 11.5 | Expectedness | 34 |
| 11.6 | Safety Monitoring Committee | 34 |
| 11.7 | Safety for PICSO | 35 |
| 11.8 | Safety for CMR | 35 |
| 11.9 | Safety of cardiac physiological measurements | 35 |
| 11.10 | Safety of blood sampling | 36 |
| 12 | STATISTICS | 36 |
| 12.1 N | Number of Participants | 36 |
| 12.2 A | nalysis of Endpoints | 37 |
| 13 | DATA MANAGEMENT | 38 |
| 13.1 | Source Data | 38 |
| 13.2 | Access to Data | 38 |
| 13.3 | Data Recording and Record Keeping | 39 |
| 14 | QUALITY ASSURANCE PROCEDURES | 39 |
| 15 | SERIOUS BREACHES | 39 |
| 16 | ETHICAL AND REGULATORY CONSIDERATIONS | 40 |
| 16.1 S | pecific Ethical Considerations for participants in emergency situations | 40 |
| 16.2 P | ossible risks and/or discomfort for patient | 40 |
| 16.3 C | Collaboration and Partnership with Commercial Companies | 40 |
| 16.4 F | easibility | 41 |
| 16.4 | .1 Facility | 41 |
| 16.5 | Declaration of Helsinki | 41 |
| 16.6 | ICH Guidelines for Good Clinical Practice | 41 |
| 16.7 | Medical Device regulations | 41 |
| 16.8 | Approvals | 41 |
| 16.9 | Reporting | 42 |
| 16.10 | Participant Confidentiality | 42 |
| 16.11 | Potential Benefits | 42 |
| 17 | FINANCE AND INSURANCE | 43 |
| 17.1 | Funding | 43 |
| 17.2 | Insurance | 43 |
| 18 | PUBLICATION POLICY | 43 |

| 19 | REFERENCES | 43 |
|----|------------|----|
| 20 | APPENDIX A | 46 |
| 21 | ADDENINY R | 17 |
| 21 | APPENDIX B | |

## 1. KEY TRIAL CONTACTS

| Chief Investigator | Prof Adrian P. Banning |
|--------------------|---------------------------------------|
| | Department of Cardiology |
| | John Radcliffe Hospital |
| | Headington, Oxford, OX39DU |
| | Adrian.Banning@ouh.nhs.uk |
| | Tel: 01865 228934 |
| | Fax: 01865 220585 |
| Sponsor | Oxford University Hospitals NHS Trust |
| Statistician | Roger Kessels |
| | Miracor Medical System |
| | Gumpendorferstrasse 109, top1.05 |
| | Austria |
| | rkessels@miricormedical.com |
| | Tel: 0031 6117175890 |
| | Tel: 0031 6117175890 |

# 2. SYNOPSIS

| Trial Title | Oxford Acute Myocardial Infarction - Pressure-controlled Intermittent Coronary Sinus Occlusion in STEMI |
|---|---|
| Internal ref. no. (or short title) | OxAMI-PICSO |
| Clinical Phase | II |
| Trial Design | Prospective single centre observational cohort study |

| Trial Participants | Patients admitted for primary percutaneous coronary intervention for ST elevation myocardial infarction | |
|---|---|---|
| Planned Sample Size | 75 patients | |
| Treatment duration | Maximum of 90 minutes | |
| Follow up duration | 6 months | |
| Planned Trial Period | 18 months | |
| | Objectives | Outcome Measures/Endpoints |
| Primary | To evaluate the effect of pressure intermittent controlled coronary sinus occlusion on the indexes of coronary physiology and on infarct size in STEMI patients at short and mid term follow up. | To evaluate the effect of pressure intermittent controlled coronary sinus occlusion on infarct size measured at cardiac magnetic resonance after 24-48 hours from revascularization. |
| Secondary | To evaluate the utility of individual biomarkers (blood components derived substances from cells, DNA, plasma etc) in the assessment of coronary artery disease and myocardial infarction investigating also how these individual biomarkers may be modified by PICSO treatment. | To evaluate the effect of pressure intermittent controlled coronary sinus occlusion on humoral biomarkers and on the evolution of parameters of coronary physiology at 24 hours and infarct size, microvascular obstruction at cardiac magnetic resonance after 6 months from revascularization. |
| Safety Endpoint | To evaluate the rate of PICSO failure deployment, coronary sinus complications, and additional time and radiation exposure associated to for PICSO deployment | |
| Device name | Pressure intermittent controlled co | ronary sinus occlusion (PICSO) |
| Device Manufacturer | Miracor Medical System | |
| Device Classification | Interventional Cardiology | |

| Protocol version no. | Effective<br>Date | Significant Changes | Previous<br>protocol<br>version no. |
|---|---|---|---|
| 2.0 | 01.04.2015 | Clarification of follow up duration Clarification for what group of patient CMR follow up is meant | v1.0 13.02.2015 |
| 3.0 | 20.06.2016 | - Extension of sample size to 75 patients to achieve a minimum of 25 patients with complete dataset | v2.0 01.04.2015 |

| Protocol version no. | Effective<br>Date | Significant Changes | Previous<br>protocol<br>version no. |
|---|---|---|---|
| 4.0 | 06.05.2016 | - Change in information about regulatory status of PICSO technology from CE-marked to non non-CE mark - Extension of recruitment beyond the period specified in the IRAS application form | V3.0 20.06.2016 |
| 5.0 | 26.02.2018 | - Extension of recruitment beyond the period specified in the IRAS application form - Extension of inclusion criteria to allow enrolment of all patients with ST elevation myocardial infarction, irrespectively of the coronary location of the culprit lesion | V4.0 06.05.2016 |

# 3. ABBREVIATIONS

| AE | Adverse event |
|----------|------------------------------------------------------------------|
| AR | Adverse reaction |
| CFR | Coronary flow reserve |
| CI | Chief Investigator |
| CMR | Cardiac magnetic resonance |
| CRA | Clinical Research Associate (Monitor) |
| CRF | Case Report Form |
| CRO | Contract Research Organisation |
| СТ | Clinical Trials |
| DMC/DMSC | Data Monitoring Committee / Data Monitoring and Safety Committee |
| FFR | Fractional flow reserve |
| GCP | Good Clinical Practice |
| GP | General Practitioner |
| ICF | Informed Consent Form |
| ICH | International Conference of Harmonisation |
| IMR | Index microrcirculatory resistance |
| IRB | Independent Review Board |

| МІ | Myocardial infarction |
|---|---|
| NHS | National Health Service |
| NRES | National Research Ethics Service |
| PCI | Percutaneous coronary intervention |
| PI | Principal Investigator |
| PICSO | Pressure controlled intermittent coronary sinus occlsuion |
| PIL | Participant/ Patient Information Leaflet |
| R&D | NHS Trust R&D Department |
| REC | Research Ethics Committee |
| SAE | Serious Adverse Event |
| SAR | Serious Adverse Reaction |
| SDV | Source Data Verification |
| SOP | Standard Operating Procedure |
| SUSAR | Suspected Unexpected Serious Adverse Reactions |
| TMF | Trial Master File |
| TSG | Oxford University Hospitals Trust / University of Oxford Trials Safety Group |

# 4. BACKGROUND AND RATIONALE

Restoration of blood flow in the infarct related artery (IRA) is the cornerstone for the current treatment of ST elevation myocardial infarction (STEMI) [1]. However in a variable proportion of patients, ranging from 30 to 40%, myocardial reperfusion is impaired, despite the apparent successful achievement of epicardial coronary artery patency [2]. This condition, known as no reflow, is due to microvasculature dysfunction and/or obstruction and it is the result of the interaction of several pathophysiological mechanisms including ischemia injury, reperfusion injury, distal embolization and tissue oedema [3].

## 4.1 Diagnosis of no reflow

Identification of no reflow and microvascular obstruction can be obtained by application of different diagnostic tools. So far cardiac magnetic resonance (CMR) represents the gold standard for detection and quantification of myocardial damage and microvascular impairment [4]. Parameters easily derived from

CMR such as infarct size, area at risk, myocardial salvage and microvascular obstruction have been shown

to be related to long term outcome.

A major limitation of CMR is the time-delay from percutaneous coronary intervention (PCI), being applied

at the earliest at the end of the revascularization procedure [4]. Early identification of patients at higher

risk of no reflow, during the PCI procedure, would be extremely useful and in such regard parameters of

coronary physiology may have a role. Indeed, measurements of blood flow and coronary microcirculation

function are now used in the catheter lab during routine PCI, using standard techniques (a pressure wire)

that are incorporated into the PCI procedure itself (by replacing the PCI procedure wire with a pressure

wire). An example of this is the measurement of the index of microcirculatory resistance (IMR), defined as

distal coronary pressure divided by the inverse of the hyperaemic mean transit time (a correlate to

absolute flow). It is measured simultaneously with the coronary pressure wire and it evaluates

microvascular resistance, independently of epicardial stenosis [5]. IMR has become the catheter-based

method of choice to independently assess coronary microcirculation [5-6]. Recent data suggest that IMR,

measured acutely in patients with MI undergoing emergency PCI, provides useful prognostic information

[7]. Specifically, a postprocedure IMR> 40 has been shown to be significantly associated with a worst long

term prognosis in terms of cardiac death and re-hospitalization for heart failure [8].

We have conducted a preliminary study, in the setting of the Oxford Acute Myocardial Infarction (OxAMI)

project, to understand the procedural aspects at PCI that may directly influence the microcirculation. The

key findings are that:

1. Coronary stenting itself reduces IMR and is thus beneficial in terms of the microcirculation.

2. Patients with a low pre-stenting IMR tend to do have little change in IMR.

3. Conversely the reduction in IMR is largest in those with a higher IMR (> 40) before stenting

4. However, a proportion of patients with high IMR can continue to have a still high (> 40) or even

further increased poststenting IMR.

Medical Device Clinical Investigation Protocol Template version DRAFT

© Copyright: The University of Oxford and Oxford University Hospitals NHS Trust 2014


26 February 2018 Version 5.0

This suggests that patients with a high pre-stenting IMR are at especially higher risk and may benefit from

additional interventions.

4.2 Retroperfusion strategy and PICSO

So far many strategies have been proposed in order to prevent and/or to treat no reflow, but none have

demonstrated a consistent beneficial effect. A new proposed approach being investigated is the

retroreperfusion strategy [9] based on the principle that it is possible to reduce the ongoing ischemia by

perfusing the myocardium through the coronary sinus.

The concept of retroperfusion is 100 years old it has been initially discarded after the advent of coronary

artery bypass grafting and PCI. Different techniques of retroperfusion are available: intermittent coronary

sinus occlusion (ICSO), synchronized retrograde perfusion (SRP) and simplified retroperfusion (SR) [10-13].

The common denominator is the temporal increase in coronary sinus pressure through the coronary sinus

occlusion (ICSO) or retroperfusion with arterial blood (SRP and SR).

PICSO is a modification of the original time-dependent ICSO and it is applied through a dedicated catheter

(PICSO Impulse catheter, Mirarcor Medical System GmbH, Vienna, Austria).

The catheter presents a balloon at the distal end. The balloon inflates and deflates cyclically once deployed

in the coronary sinus, leading to intermitted coronary sinus pressure increase. This intermittent increase

in coronary sinus pressure leads to an improved perfusion of the ischemic area with potential benefit in

terms of myocardial salvage through 3 mechanisms: 1) redistribution of blood flow from the remote

myocardium to the border zone of the ischemic myocardium [14]; 2) enhanced wash out of noxious,

inflammatory factors and embolic material across the microvascular bed (suction effect upon balloon

release) [15]; 3) improvement in collaterals through release of vascular growth factors as consequence of

venous pressure increase [16-17].

The PICSO technology has revealed to be effective in several models by reducing infarct size (IS) [18] and

a metanalysis on seven studies on animal models has confirmed a statistically significant -29% (CI95% -

40.9 – -17.7, p<0.001) reduction in IS compared to control group [19]. Moreover, it has also been shown

that the benefit from PICSO treatment is directly proportional to the pressure reached in the coronary

sinus during the balloon inflation and thus to the increase in coronary wedge (CW) pressure, which is the

pressure associated to the blood flow provided to the ischemic region by collateral branches [20].

The Prepare-PICSO study represents the first-in-man experience with the PICSO device [21]. On a small

sample of 15 patients with stable angina the PICSO treatment showed to be firstly safe and, as observed

in the animal models, was associated to a significantly increase in coronary sinus pressure as well in mean

CW pressure in the distal left anterior descending (LAD) coronary artery [21].

These findings have triggered the Prepare-RAMSES study in which PICSO treatment was investigated for

the first time in man in patients with STEMI [22]. The results of the study have been recently published.

The study was initially designed to include 30 patients with anterior STEMI with PICSO treatment for 90

minutes after the completion of primary percutaneous coronary intervention (PPCI). The study enrolled

only anterior STEMI since expected to be responsive to the PICSO device, being mainly the anterior wall of

the myocardium drained by the coronary sinus. The device resulted to be safe, with a median implantation

time of 12 minutes. The primary endpoint was the reduction in IS at cardiac magnetic resonance (CMR) at

2-4 days and 4 months. The PICSO group was compared with a matched control group of patients.

Although the study did not show an overall difference in the reduction in IS in the PICSO group [22], IS

reduction appeared to be significantly related to the quantity of PICSO treatment (pressure achieved in

the coronary sinus x time of treatment) and significantly higher in the small subgroup of patients receiving

high PICSO quantity.

It is possible that the study did not reach the primary endpoint due to some limitations in its design. First

of all the small sample size has to be acknowledged, since the investigators managed to fully deliver the

PICSO treatment only to 12 patients (63% of the initially intended sample size). Moreover, the study

presented a potential "selection bias" that drove the investigators to include in the study "relatively healthier" patients in which anticipated benefit was limited: 40% of patients enrolled presented with a Thrombolysis In Myocardial Infarction (TIMI) flow > 1, e.g. presented with an open coronary artery at the time of primary PCI. Moreover the application of PICSO treatment at the end of the PPCI may have blunted the expected benefit: the device was deployed after stenting, the stage the procedure known to be at higher risk of distal embolization of atherothrombotic debris downstream the coronary microvasculature [22].

Identification of "higher risk" STEMI patients is thus crucial in order to confirm a clear benefit associated to the PICSO device.

### 4.3 Study Hypothesis

The Oxford Acute Myocardial Infarction - Pressure-controlled Intermittent Coronary Sinus Occlusion in STEMI (OxAMI-PICSO) study aims to analyze the potential benefit of PICSO in a selected population of STEMI patients. In patients with prestenting high IMR, and thus with larger infarct size and more compromised microvasculature status, PICSO treatment added to the conventional revascularization gold standard is expected to be associated to a better myocardial reperfusion. This will be assessed by measurement of indexes of coronary physiology and by CMR evaluation of indexes associated to infarct size, myocardial salvage and microvascular obstruction, and other biomarkers. The comparator group will be matched participants previously enrolled in the OxAMI study, with STEMI and with a prestenting IMR above 40.

### 5. OBJECTIVES AND OUTCOME MEASURES/ENDPOINTS

| Objectives | Outcome Measures/Endpoints |
|------------|----------------------------|

## **Primary Objective**

To assess the impact of PICSO on coronary physiology parameters, on infarct size, on myocardial salvage and on microvascular obstruction at CMR in a selected population of STEMI patients at higher risk of no reflow and with the theoretical prerequisites that make more likely to respond to PICSO treatment. The control group will be represented by a highly matched group of patients from the ongoing Ox-AMI (Oxford Acute Myocardial Infarction) project (Ethics Ref 11/SC/0397), who have undergone all other aspects of the study protocol, including assessment of coronary physiology at 24 hours post primary PCI, 24-48 hours and 6 months CMR, but who have not received PICSO treatment.

Area at risk, Infarct size, Myocardial salvage and microvascular obstruction measured by cardiac magnetic resonance at 24-48 hours

#### **Secondary Objectives**

The OxAMI-PICSO study aims to evaluate the utility of individual biomarkers (blood components derived substances from cells, DNA, plasma etc) in the assessment of coronary artery disease and myocardial infarction. The OxAMI-PICSO may show also how these individual biomarkers may be modified by PICSO treatment.

Coronary flow reserve (CFR), Fractional Flow reserve (FFR), index of microcirculatory resistance (IMR) measured at 24 hours after PCI.

Infarct size and microvascular obstruction extent measured by cardiac magnetic resonance at 6 months

Individual Biomarkers related to coronary artery disease/myocardial infarction at three time points (PCI, 24/48 hours after PCI and 6 months). These include: blood biomarkers of myocardial injury, metabolism and inflammation.

#### **Tertiary Objectives**

To evaluate the rate of PICSO failure deployment, coronary sinus complications, and additional time and radiation exposure associated to for PICSO deployment

Rate of PICSO failure deployment

Rate of coronary sinus complications: perforation, dissection, thrombosis

Time for PICSO deployment / additional screening time and radiation dose

#### 6. TRIAL DESIGN

The OxAMI-PICSO study is a prospective single centre observational cohort study of the use of PICSO in patients presenting for primary PCI for acute myocardial infarction. The OxAMI- PICSO study is based upon the established framework of the OxAMI study (Ethics Ref 11/SC/0397).

26 February 2018 Version 5.0

Patients, age 30-90, presenting with ST elevation myocardial infarction will be considered for inclusion in

the study. Measurement of IMR before stenting is an essential prerequisite for the study: only patients

with pre-stenting IMR > 40 will be considered eligible for the PICSO treatment. Patients with IMR≤ 40 will

remain in the study but will not undergo PICSO treatment. The procedure for consent in patients

undergoing emergency PCI will be as already established in the ongoing OxAMI study, and is discussed

below in Section 8.1.2.

The PCI procedure will be undertaken in a standard fashion, and include the use of pressure wire

measurements before and after stent deployment. Aspiration or distal protection devices may be used if

clinically indicated and where vessel anatomy is suitable. The devices used and the procedural techniques

will be driven by clinical decision making at the patient and institutional level, and carried out in

accordance with the Oxford University Hospitals NHS Trust (OUHT) departmental guidelines for PCI.

PICSO treatment will be added on top of the conventional treatment.

The protocol will constitute of 5 main stages described in details in the next sections (Section 8.3).

Only patients with pre-stenting IMR > 40 and who assent to receive PICSO treatment will undergo 24 hours

coronary angiogram with coronary physiology measurement, 24-48 hours CMR scan and 6 months CMR

scan. Patients who assent to participate in the study but in whom the prestenting IMR ≤ 40, or those in

whom the prestenting IMR > 40 but the participant declines PICSO treatment will remain in the study for

blood sampling and clinical data collection at the same follow up time points (24 hours, 48 hours and 6

months). A summary of the study design, indicating the time points and procedures, is shown in Section

8.3.

7. PARTICIPANT IDENTIFICATION

7.1. Trial Participants

Participants aged 30-90 years old, referred for emergency diagnostic coronary angiography presenting with ST elevation myocardial infarction, with the intention to proceed to primary PCI with stenting.

#### 7.2. Inclusion Criteria

Participants must satisfy the following conditions:

- Male or Female, aged 30 to 90 years,
- Clinical presentation with STEMI
- Referred for coronary angiography with view to proceed to PCI with stenting.

#### 7.3. Exclusion Criteria

The participant may not enter the study if ANY of the following are known to apply:

- Patients in whom safety or clinical concerns preclude participation.
- Known anaemia (Hb <9).
- Pregnant or breast feeding females.
- Revascularization by mean of balloon angioplasty without stenting
- History of stroke, TIA or reversible ischemic neurological disease within last 6 months
- Known severe renal failure (eGFR < 30 ml/min/1.73m2) or history of dialysis or renal transplant
- Previous coronary bypass artery grafting
- Known severe valvular abnormalities
- Previous STEMI presentation
- Presentation with cardiogenic shock
- Severe bradycardia (Heart rate < 50 beats per minutes)</li>
- STEMI due to stent thrombosis
- Unconscious on presentation

- Non-cardiac comorbidities and life expectancy < 1 year</li>
- Use of warfarin
- Presence of pacemaker or other electrodes in the coronary sinus
- Contraindications to adenosine
- Additional exclusion criteria for participants undergoing CMR
- claustrophobia which limits / prevents participants from remaining in CMR scanner.
- o patients who cannot lie flat on the scan table.
- patients with metallic implants, pacemakers, implantable defibrillators etc, unless known to be
   CMR compatible.
- o patients with known allergy to medium of contrast (gadolinium)

#### 8. TRIAL PROCEDURES

#### 8.1. Informed Consent

Informed consent will be obtained, with the recruitment approach to the patient, as described below.

#### 8.1.1 Patients proceeding to emergency angiogram/PCI

The clinical treatment of these patients is in the emergency context and delays to treatment are detrimental. It is necessary to administer prompt emergency treatment and it is not always possible to identify and approach a Consultee beforehand. Thus we would seek a waiver, as described in Section 32(9) of the Mental Capacity Act, since

- a) the treatment needs to be given urgently,
- b) it is necessary to take the action for the purpose of the research urgently,

but

c) it is not reasonably practicable to consult prior to enrolling the patient.

In this situation the Mental Capacity Act allows the participant to be enrolled with a agreement of a

registered medical practitioner (RMP) not involved in the research or in accordance with a

procedure agreed with the appropriate body (i.e. REC). Since this is only applicable for the duration

of the emergency we will seek written informed consent as soon as reasonably practicable (see

diagram and Section 8.1.1.2 below). This process includes an important role for a healthcare

professional as a type of patient "advocate". This is discussed in section 8.1.1.2 below. We also seek

approval from the REC for the waiver procedure.

8.1.1.1 Verbal assent

Because of the urgency of the situation it is not feasible to obtain fully informed written consent.

Fully informed consent requires that the potential participant have time to read and reflect on a

patient information sheet which in this context is clinically inadvisable. We therefore propose to

obtain verbal assent so as to optimize the amount of appropriate information conveyed to potential

participants acutely and minimize the clinical risks involved with substantial delay. The research

study will be discussed verbally with the patient and the risks and benefits explained.

In detail the patient at the time of verbal assent process will be informed that as part of the research

project he might undergo to some extra blood samples and to measurement of the index of

microcirculatory resistance (IMR) which allows to have an indirect assessment of the entity of the

ongoing heart attack. The patient will be also informed that in case IMR value will be greater than

40, thus suggesting a possible significant damage to the heart muscle that may benefit from

additional treatment, he might be asked to provide assent for PICSO treatment. Patients with pre-

stenting IMR ≤ 40 or those with prestenting IMR > 40 who elect not to receive PICSO treatment will

be given the opportunity to continue to participate within the OxAMI-PICSO study, but without the

use of the PICSO device.

Medical Device Clinical Investigation Protocol Template version DRAFT

© Copyright: The University of Oxford and Oxford University Hospitals NHS Trust 2014


Participants will be reminded that they have the right to withdraw from the study at any stage and that this will not affect their treatment or human rights. The research and clinical team have extensive experience of patient assent, and the role of a Patient Advocate (see below), through the recruitment of approximately 250 participants undergoing emergency PCI for STEMI in the OxAMI study.

Only conscious patients, able to provide verbal assent will be enrolled in the study.

#### 8.1.1.2 Patient Advocate

Because of the urgency of the situation it is not feasible to consult prior to enrolment, a RMP or patient "advocate" will be identified to act in accordance with 32(9). The Patient Advocate will act as witness and documenter of the verbal consent process for all conscious potential participants and/or overseer of the waiver process (8.1.2.3) as a whole. This RMP will be present at the time of emergency treatment, but is not part of the research team. The Advocate will ensure that the verbal consent process is undertaken, that the patient does not object (i.e. the patient "assents" rather than "dissents"), and that the researcher has taken practical steps to explain the study, risks and benefits, within the context of the emergency clinical situation, and in accordance with the clinical status of the patient. The Advocate in this situation will be a healthcare professional such as a specialist nurse. Assessment of patients in this context is within their professional capacity and the role here will be to witness verbal consent or assent.

Most of the nursing staff attended a series of seminars to make them aware of their specific roles and responsibilities in this situation, and they have acted as patients' advocates through the recruitment of approximately 250 participants undergoing emergency PCI for STEMI in the ongoing OxAMI study. These seminars have been directed by an ethicist who is not directly involved with the research project. We will continue to provide this training and draw on the extensive experience of the members of the clinical team currently acting as a Patient Advocate.



### 8.1.1.3 Post-emergency phase

Once the emergency phase is over and treatment has been delivered, we will seek full written informed consent as soon as practical. For most patients this means within 12 hours of admission.

This consent will be a two parts process:

- a) We will seek consent to allow use of data and samples already acquired during the emergency phase
- b) We will seek consent for ongoing participation in the study.

If the participant elects to withdraw from the study at this point then we will seek consent to use the data and samples already acquired. If this is not given, then all research data and samples acquired during the emergency treatment will be destroyed, otherwise only data acquired in the emergency situation will be retained in the study.

If a patient is unable to provide informed consent at this stage due to deterioration in clinical condition, we propose to keep the data and samples acquired under the assent phase. We would not seek further 'consent' from relatives at the risk of causing undue distress.

# 8.2. Discontinuation/Withdrawal of Participants from Trial Treatment

## 8.2.1 Study Withdrawal

We anticipate and have made provision for withdrawal when the emergency exception period is complete; if a patient is assessed and has capacity then they may completely or partially withdraw at any time. This possibility will be made clear as a part of seeking of full written informed consent after the initial emergency procedure.

### 8.2.2 Participant death:

If the participant dies before giving full written consent then we propose to continue using the data and samples obtained. We would not seek further 'consent' from relatives at the risk of causing undue distress.

## 8.3 Study timeline (see "Integrated flowchart for OxAMI-PICSO study" as below)

The OxAMI-PICSO study will take place beside an ongoing large prospective observational study in STEMI patients (OxAMI study). Patients fulfilling the OxAMI-PICSO criteria will be invited to participate in the study. OxAMI-PICSO study will constitute of 5 main stages:



# 8.3.1 Stage 1: Pre-Stenting

- 1. Diagnostic angiography will be performed in the standard manner using appropriate catheters.
- 2. Bivalirudin will be administered (0.75mg/kg bolus followed by an infusion of 1.75 mg/kg/min for up 4 hours after the procedure as clinically warranted), as routinely used for PCI. The lesion will be

crossed with a coronary guide wire in the usual manner for PCI. Normal blood flow will be rapidly

achieved by thrombus aspiration and/or predilation

3. Pre-stenting coronary physiology parameters, namely FFR, CFR and IMR, will be measured, using

a pressure wire, as used for routine clinical measurements in patients undergoing PCI.

4. If pre-stenting IMR is > 40, patients will be invited to receive the PICSO device. If pre-stenting IMR

is ≤ 40 PICSO device will not be proposed, but the patient will be invited to remain in the study for

serial blood sampling (procedural-6 hours-24 hours and 48 hours) and routine clinical data

collection.

8.3.2 Stage 2: PICSO treatment

1. In patients with IMR >40 who assent to PICSO treatment, the PICSO device will be deployed as

already previously described in the literature [22] (Section 9.2). The overall duration of PICSO will

be no less of 60 minutes up to a maximum of 90 minutes in order to ensure a PICSO delivery dose

of 800 mmHg.

8.3.3 Stage 3: Stenting

1. Stenting is performed as usual clinical practice.

2. Post-dilation is left to operator's discretion, as in clinical routine.

3. At the end of the procedure a final reassessment of coronary physiology parameters is performed

again as previously described.

Blood samples may be taken, (by 5 or 10 ml syringes), at the following time-points, from both

peripheral vein (V), using the venous cannula, from the coronary sinus (CS) using a CS sampling

catheter, or the PICSO delivery sheath, and from the coronary artery (C) either via the guide catheter

used for the procedure or an aspiration catheter placed through the guide catheter:

Sampling point (1): beginning of procedure V, C

Sampling point (2): placement of PICSO device V, CS, C

Sampling point (3): end of procedure V, CS, C

Sampling point (4): end of PICSO treatment period V, CS,

Sampling point (5): 6 hours after 1<sup>st</sup> stent deployment

For patients in whom an aspiration catheter or protection device is used during PCI, blood, thrombus and/or atheromatous plaque material may be retrieved during the procedure. These materials, which are usually discarded, will be retained for analysis. Data on the PCI procedure and any device or technology used will be collected.

# 8.3.4 Stage 4: 24-48 hours post PCI

Full written consent to take part to the OxAMI-PICSO study is obtained as soon as practicable. The following study assessments may be carried out:

- Repeat coronary angiogram for assessment of coronary physiology parameters assessment –
   for participants who receive the PICSO device only
- 2. Cardiac magnetic resonance for participants who receive the PICSO device only
- 3. Venous blood sampling for biomarker measurement
- 4. Data Collection, Patient Reported Outcomes and Cardiovascular Outcomes

## 8.3.5 Stage 5: 6 months post PCI

Participants will be invited to attend the hospital as an outpatient at approximately 6 months post-PPCI for the following research assessments

- 1. Cardiovascular MRI for participants who receive the PICSO device only
- 2. Blood sampling for biomarker measurement
- 3. Data Collection, Patient Reported Outcomes and Cardiovascular Outcomes

8.4 Definition of End of Trial

Recruitment to the study will cease as soon as 25 participants have undergone PICSO treatment and have

completed follow-up at 6 months. The study will end on the date of the last CMR at 6 months follow up of

the last participant recruited.

9. STUDY ASSESSMENT

9.1 Data Collection, Patient Reported Outcomes and Cardiovascular Outcomes

Data on the clinical procedures and any devices and/or imaging technologies used will be collected.

Medical history will be taken from the patient once informed consent has been given and relevant sections

of the medical notes may be accessed by the study team. Clinical outcomes and MACE will be ascertained

during the follow-up appointment with the patient, by accessing relevant sections of the medical notes,

ONS database and existing databases of cardiac outcomes and treatment (such as the CCAD and MINAP

databases), or by contacting the GP if appropriate.

9.2 PICSO device

See Section 10

9.3 Analysis of CMR

Cardiac related parameters will be derived for further analysis. Analyses will be performed according to

published methods and will be focused on the assessment of different cardiac components including

anatomy, function, tissue, flow and metabolism (i.e. ventricular volumes, wall motion, infarct size, area at

risk, myocardial salvage and microvascular obstruction) [23]. These parameters are partly used both

clinically and in research settings (e.g. heart volumes, myocardial mass).

9.4 Analysis of cardiac physiological measurements

Cardiac and/or coronary flow and pressures will be measured, before and after stenting and during the

repeat coronary angiogram at 24 hours post-PPCI, using commercially available measurement guidewires

according to standard techniques that are in routine use in current PCI practice. The guidewire contains a pressure-temperature sensor to allow for calculation of the physiological parameters. The guide wire is calibrated at the beginning of the PCI and then advanced into the distal third of the culprit artery. Calculations will be based on measurements of proximal and distal coronary pressure(s) and mean transit time (in seconds) during maximal hyperemia, as previously described. Briefly a pressure wire (Radi; St Jude Medical, St Paul, MN, USA) is placed in the LAD distal to the lesion. Baseline mean aortic pressure (Pa), mean distal pressure (Pd) and Pd/Pa ratio will be recorded. Thermodilution-based measurement of CFR and IMR will be performed by injecting in the IRA 5 ml of room temperature saline solution and recording mean transit time (meanTt) at baseline and after induction of maximal hyperaemia by intravenous infusion at a rate of at a rate of 140 mg/kg/min. Once hyperaemia is achieved the following parameters will be obtained: FFR (Pd/Pa during hyperemia), CFR (meanTtbaseline/meanTthyperaemia) and IMR (Pdhyperaemia\* meanTthyperaemia).

## 9.5 Analysis of blood samples

Blood samples collected at the respective time points will be prepared under standard laboratory protocols, blood and its derived components will be aliquoted and stored, as necessary, in appropriate conditions for further analyses. The samples will be analysed for known and novel biomarkers related to coronary artery disease and myocardial infarction, using techniques such as enzyme immunoassay, flow cytometry etc. Samples may be assayed using novel platforms to investigate the potential utility against the existing techniques. Samples may be stored and sent to other centres, outside the UK, for specific analyses, according to the availability of specialist techniques. Depending on specific informed consent being given by participants, blood will be stored for DNA extraction and future genetic analysis, including typing of SNPs and for whole genome analysis. Specific genetic variants may be used to guide invitations to participate in future studies.

### 9.6 Analysis of particulate debris

Intracoronary thrombus / plaque material obtained with the use of thrombus aspiration at any stage of the procedure will be prepared under standard laboratory protocols and stored at -80°C for further analyses. Snap frozen debris may be analysed using immunohistochemical stains, including antibodies to CD68, smooth muscle actin, CD3, and CD20, Tissue Factor [24], Vascular Endothelial Growth Factor (VEGF) [25], MMPs 2 and 9 [26], cellular proliferation and apoptosis [27-29]. Samples may also be analysed by extraction of mRNA for RT-PCR, or for levels of proteins/lipids using proteomics/lipidomics approach or other molecular markers using novel technologies.

### 10. IDENTIFICATION & DESCRIPTION OF THE INVESTIGATIONAL DEVICE

### 10.1 Device description

The PICSO Impulse System consists of the PICSO Impulse console (101.100.000.000) and PICSO impulse catheter (300.100.000.010) by Miracor Medical Systems (Gumpendorferstrasse 139, Top1.05 Vienna, A-1060).







PICSO Impulse Catheter

Each PICSO Impulse catheter will have a serial number, which will be recorded for traceability during and after completion of the study.

The PICSO Impulse catheter presents a balloon at the distal end. The balloon inflates and deflates cyclically once deployed in the coronary sinus, leading to intermitted coronary sinus pressure increase. This intermittent increase in coronary sinus pressure leads to an improved perfusion of the ischemic

area with potential benefit in terms of myocardial salvage through 3 mechanisms: 1) redistribution of

blood flow from the remote myocardium to the border zone of the ischemic myocardium [14]; 2)

enhanced wash out of noxious, inflammatory factors and embolic material across the microvascular

bed (suction effect upon balloon release) [15]; 3) improvement in collaterals through release of vascular

growth factors as consequence of venous pressure increase [16-17].

The PICSO Impulse catheter is a 8F double lumen catheter with a 15.5x20mm long balloon at the distal

end. The catheter is connected to the console through two pneumatic tubes in which helium is shuttled

to and from the balloon. In addition, the coronary sinus pressure is monitored through the center lumen

of the catheter. The catheter is placed in the coronary sinus over a 0.025' wire by a 8.5Fr pre-shaped

delivery long steerable sheath (Oscor Destino Steerable Sheath DS856750/22) inserted in the femoral

vein. Femoral vein access is obtained as routine practice according to Seldinger technique. Once the

catheter is placed, the guidewire is removed and the steerable sheath is retracted in the right atrium

for support. PICSO deployment median time has been estimated to be of 12 minutes (Interquartile

Range 9-18 minutes)

The PICSO Impulse Catheter is then connected to the PICSO Impulse console. The PICSO Impulse

Console automatically operates the PICSO Impulse Catheter. The balloon is intermittently inflated and

deflated using helium, based on coronary sinus pressure and synchronized with the ECG. The monitor

displays the inflation/ deflation state of the balloon, as well as trend graphs and time counters; Live

graphs display curves and numeric values of ECG, coronary sinus pressure, aortic pressure and auxiliary

input. It is easy to use and provides direct feedback on the patient's individual therapy using the 'PICSO

Dose', which is defined as the sum of the coronary sinus pressure modulation for all PICSO cycles

applied. All data are automatically stored and can be retrieved for later analysis for each patient. The

unit is transportable and runs on battery supply if needed during patient transportation.

Once the PICSO Impulse catheter is connected to the consoled, by activating the "START" button, the

distal balloon will be cyclically inflated. Each cycle starts with a balloon inflation triggered by QRS

Medical Device Clinical Investigation Protocol Template version DRAFT

© Copyright: The University of Oxford and Oxford University Hospitals NHS Trust 2014

complex on ECG monitoring. During balloon inflation coronary sinus pressure will progressively increase

till reaching a plateau, then coronary sinus occlusion is stopped by balloon deflation. For security, each

balloon inflation has a maximum limit of 30 seconds in duration. The deflation interval between two

cycles has a minimum duration of 3 seconds.

In the OxAMI-PICSO the PICSO Impulse system will be adopted in a highly selected population of

patients with ST elevation myocardial infarction, characterized by a possibly impaired microvasculature

impairment at the time of the PCI, as expressed by a prestenting elevated index of microcirculatory

resistance (> 40). The aim is to assess the extent of infarct size after 24-48 hours in such specific group

of patients. Propensity-score matched historical patients from the ongoing OxAMI study will be controls

in the OxAMI-PICSO study.

All the investigators using the PICSO device will undergo a specialist training programme completion,

including the performance of the first cases under the supervision of a proctor expert. Educational

training sessions for use of the PICSO will be provided to all clinical staff (nurses, radiographers,

physiologists) involved in the care of patients who have received PICSO.

**10.2 Device Safety** 

PICSO treatment is safe. Potential complications associated to PICSO may include:

a) Bleeding due to damage to the coronary sinus where the PICSO catheter is placed

b) Bleeding in the groin from the femoral vein access.

c) Long term blockage of the coronary sinus where the PICSO catheter sits.

d) Helium leak from the catheter into the blood. A leak of helium into the patient could occur with a

balloon rupture or hole. However the risk is significantly mitigated since the system can automatically

detect any leakage and stop the procedure. The maximum helium volume that could enter the patient

using the PICSO system is less than 10 ml. This volume is approximately 1/3 of the volume that could

leak from a bursting intra-aortic balloon pump (IABP) catheter, that are used in routine clinical practice

in the aorta (i.e arterial circulation), whereas the PICSO catheter is used exclusively in the venous

Medical Device Clinical Investigation Protocol Template version DRAFT

© Copyright: The University of Oxford and Oxford University Hospitals NHS Trust 2014


circulation.. A helium leak from the PICSO system is therefore regarded to constitute a low risk to the

patient.

Data about PICSO are continuously increasing and in the two main studies performed in man so far

(PREPARE-PICSO and PREPARE-RAMSES) only one procedure adverse event (tamponade secondary to

coronary sinus perforation) has been described. This rate (<3%) of complication is further lower than

that associated to the routine elective electrophysiological procedures to the coronary sinus in the

context of tachycardia ablation or cardiac resynchronization therapy.

It is possible that the PICSO balloon may be dislodged from the coronary sinus into the right atrium.

This event has no known safety implications for the patients, but it may affect the efficacy of the PICSO

treatment. The PICSO console will detect the occurrence of such event and alert the clinical team. In

such a scenario balloon repositioning will only be considered if the treatment time-interval is less than

60 minutes. In order to minimize the risk for the patient, repositioning will be performed under

fluoroscopic guidance in the catheterization laboratory. Once the balloon is repositioned, the PICSO

treatment will be continued to achieve a minimum total treatment time of 60 minutes to a maximum

of 90 minutes from the time of stent deployment.

All the investigators using the PICSO device will undergo a specialist training programme completion,

including the performance of the first cases under the supervision of a proctor expert. Educational

training sessions for use of the PICSO will be provided to all clinical staff (nurses, radiographers,

physiologists) involved in the care of patients who have received PICSO. Patients undergoing PICSO

treatment will be strictly monitored, according to the standard clinical care guidelines, during and after

the PICSO treatment in order to minimize or to early detect possible issues associated to the treatment.

After the procedure, when the PICSO treatment is still ongoing, the patients will be monitored in the

Recovery Assessment Area in order to guarantee a rapid access to the Catheterization Laboratory, if

required.

The additional x-rays used for the placing of the device is extremely low in the context of the exposure

associated to the standard primary PCI procedure. The radiation dose associated with the placement

Medical Device Clinical Investigation Protocol Template version DRAFT

© Copyright: The University of Oxford and Oxford University Hospitals NHS Trust 2014

of the device is estimated to be 4.3 mSv, which is approximately equivalent to 22 months exposure to UK background radiation. This may theoretically be associated with an increased lifetime risk of developing a cancer of 0.06%. This compares with the risk of developing a cancer in the general population of around 30% to 40%. So overall this represents a very small addition to the underlying cancer risk from all causes.

The radiation exposure in case of repositioning the PICSO balloon is estimated to be less than that associated with the device implantation. Therefore patients undergoing repositioning would have a global radiation dose associated to the PICSO device of no more of 8 mSv.

# 10.3 Device Accountability

PICSO Impulse console and PICSO Impulse catheter will be provided by Miracor Medical Systems. We will be documenting the number of devices, with their lot numbers, that will be shipped to the John Radcliffe Hospital. PICSO Impulse console will be placed in the Catheterization Laboratory of the John Radcliffe Hospital, connected to electric supply in order to assure full charge of the battery. After their delivery, the PICSO Impulse catheters will be stored in the storage room of the Catheterization Laboratory f the John Radcliffe Hospitals and kept in a cool, dry place.

We will document on the CRF the LOT number and expiry date for each balloon for each patient.

### 11 SAFETY REPORTING

### 11.1 Definitions

| Adverse Event (AE) Any unto | vard medical occurrence, unintended disease or injury or any |
|---|---|
| untoward | clinical signs (including an abnormal laboratory findings) in |
| participar | ts, users or other persons whether or not related to the |
| investigat | ional medical device. This includes events related to the |

investigational device or comparator, events related to the procedures involved (any procedure in the protocol). For users or other persons this is restricted to events related to the investigational medical device. Adverse Device effect An adverse event related to the use of an investigational medical device. (ADE) This definition includes any events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational device. This definition also includes any event resulting from user error or form intentional misuse of the investigational device. Serious Adverse Event An adverse event that: (SAE) Led to death Resulted in serious deterioration in the health of the subject that: resulted in a life-threatening illness or injury o resulted in a permanent impairment of a body structure or a body function required in-patient prolongation care or hospitalisation o resulted in medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.

This includes device deficiencies that might have led to a serious adverse event if: a) suitable action had not been taken or b) intervention had not been made or c) circumstances had been less fortunate. These are handled under the SAE reporting system. Planned hospitalisation for a pre-existing condition, or a procedure required by the trial protocol, without serious deterioration in health, is not considered a serious adverse event. Any untoward medical occurrence that can be attributed wholly or Serious Adverse Device partly to the device, which resulted in any of the characteristics of a Effect (SADE) serious adverse event as described above. Unanticipated Serious Adverse Device Effects (USADE) Any serious adverse device effect which, by its nature, incidence, severity or outcome, has not been identified Device deficiency Inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance. Device deficiencies include malfunctions, use errors and inadequate labeling. Device deficiencies that did not lead to an adverse event, but could have led to a medical occurrence if suitable action had not been taken, or intervention had not been made or if circumstances had been less fortunate

User error

Act or omission of an act that results in a different medical device response than intended by the manufacturer or expected by the user.

Use error includes slips, lapses and mistakes. An unexpected physiological response of the subject does not itself constitute a use error.

Severity definitions

The following definitions will be used to determine the severity rating for all adverse events:

Mild: awareness of signs or symptoms, that does not interfere with the subject's usual activity or is transient that resolved without treatment and with no sequelae.

Moderate: a sign or symptom, which interferes with the subject's usual activity.

Severe: incapacity with inability to do work or perform usual activities.

### 11.2 Causality

The relationship of each adverse event to the trial device may be determined by the manufacturer and/or a medically qualified Investigator according to the following definitions:

**Not related:** The event is clearly related to other factors such as the patients/participants clinical condition, therapeutic intervention, concomitant medication.

**Unlikely:** The event is probably produced by other factors such as the patients/participants clinical condition, therapeutic intervention, concomitant medication and does not follow a known response pattern to the device

**Possibly:** The event follows a reasonable temporal relationship form the time of placement/administration

and/or follows a known response pattern to the device but could have been caused by other factors such

as the patients/participants clinical condition, therapeutic intervention, concomitant medication.

Most probable: The event follows a reasonable temporal relationship form the time of

placement/administration and/or follows a known response pattern to the device and could not have been

caused by other factors such as the patients/participants clinical condition, therapeutic intervention,

concomitant medication. Further the event immediately follows the administration/placement of the

device and improves on stopping or removing the device.

11.3 Procedures for Recording Adverse Events

All adverse events (including ADEs) and device deficiencies occurring during the course of the study will be

recorded on the CRF whether or not attributed to the trial device. The information recorded will include

but not be limited to:

• A description of the event

• The dates of the onset and resolution

Action taken

Outcome

Assessment of relatedness to the device

Whether the AE is serious or not

Whether the AE arises from device deficiency

Whether the AE arises from user error

The severity of events will be assessed on the following scale: 1 = mild, 2 = moderate, 3 = severe.

AEs/ADEs considered related to the device as judged by a medically qualified investigator or the Sponsor

will be followed either until resolution, or the event is considered stable.

26 February 2018 Version 5.0

It will be left to the Investigator's clinical judgment to decide whether or not an AE/ADE is of sufficient

severity to require the participant's removal from treatment. A participant may also voluntarily withdraw

from treatment due to what he or she perceives as an intolerable AE/ADE. If either of these occurs, the

participant must undergo an end of trial assessment and be given appropriate care under medical

supervision until symptoms cease, or the condition becomes stable.

11.4Reporting Procedures for Serious Adverse Events

Reporting of all Serious Adverse Events will be done in accordance with the European Commission

Guidelines on Medical Devices Serious Adverse Event Reporting (MEDDEV 2.7/3; December 2010).

SAEs/SADEs that pose an immediate risk to patient health or safety, will be reported to the trial

DSMC/Sponsor immediately or no later than 24 hours after the Investigator is aware and to the device

manufacturer, competent authority and the REC within 2 calendar days of the Chief Investigator becoming

aware of the event.

All other reported SAEs/SADEs will be reported to the trial DSMC and Sponsor competent authority within

7 calendar days of notification, if appropriate. This will not include SAEs that may be expected as part of

the risks of routine care. Adverse device events (SADEs, USADEs) and device deficiencies will also be

reported to the device manufacturer. All SAEs will be followed up to resolution.

SAEs/SADEs will be recorded for a time period going from verbal assent/PICSO device adoption to 30 days

following the use of the device.

11.5Expectedness

Expectedness will be determined according to the Manufacturers risk analysis report

11.6Safety Monitoring Committee

The Oxford University Hospitals Trust will conduct a review of all SAEs/SADEs for the trial reported during the quarter and cumulatively. The aims of this committee include:

- To pick up any trends, such as increases in un/expected events, and take appropriate action
- To seek additional advice or information from investigators where required
- To evaluate the risk of the trial continuing and take appropriate action where necessary

# 11.7 Safety for PICSO

See 10.2

#### 11.8 Safety for CMR

CMR is a safe and non-invasive technique with no known risk when appropriately supervised. It does not involve ionising radiation. Potential participants with ferromagnetic objects in their bodies or with implanted devices which can be damaged by the CMR magnet will be excluded. All participants entering the scanner room are screened for such objects. Gadolinium contrast is widely used for clinical indications in CMR and is safe. Occasionally it may cause a mild headache, nausea, itching and very rarely (< 1 in 1000) a more severe allergic reaction. It is cleared within hours by the body. Gadolinium has recently been associated with nephrogenic systemic fibrosis in patients with severe renal dysfunction; hence, as per departmental guidelines based on Food and Drug Administration guidelines, all patients with glomerular filtration rate (GFR) < 30 ml/min (stage 3-5 renal disease) should be not be given gadolinium. Participants for whom there is a possible history of metal in the eye and we are unable to find documented clinical evidence that the metal has been removed, will be offered an orbital (eye) x-ray prior to their cardiac CMR scan to confirm or negate presence of metal in the eye. This will add 0.1 mSv additional radiation exposure; this is 1/260 of that incurred during a standard coronary angiogram procedure. There are no contraindications to short periods of supplementary oxygen in appropriately selected patients.

### 11.9 Safety of cardiac physiological measurements

Coronary pressure wire studies are routinely performed during PCI procedures. The repeat catheterizations 24-48 hours after PCI are not part of routine practice and special attention will be paid to minimize radiation and use of contrast agent. The risk of repeating cardiac catheterization is low; a commonly occurring consequence is bruising at the site of vascular access which can be treated with simple analgesia. Based on local audit data, the average radiation exposure for a patient during routine angiography is 5 mSv. The additional IMR measurement adds on average only 1.6 mSv to the procedure. The follow up visits for IMR measurement also allows a valuable clinical opportunity to assess the result of initial PCI, which not otherwise be performed.

# 11.10 Safety of blood sampling

Blood sampling performed during the procedure will be performed through either the femoral venous sheath, coronary sinus catheter or coronary artery catheter. The femoral artery sheath and coronary artery catheter are required for and routinely used for PCI to be carried out. Some discomfort and possible complications are associated with placement of the femoral arterial sheath, but this is already clinically indicated as a necessary part of the PCI. The femoral venous sheath is not routinely placed for all PCI procedures, but is used whenever additional venous access during PCI is required clinically, for example to place catheters in to the venous system, or catheters or pacing electrodes in to the right side of the heart, or infusion of drugs during the PCI procedure. Potential risks and complications associated with venous sheath placement are much less than arterial sheath placement, because blood is not under arterial pressure and because other potential risks are intrinsically lower in the venous circulation. Placement of a coronary sinus catheter is not routinely used during PCI, but is used routinely using during other commonly performed cardiac interventions. The risk of additional complications is very low. The average volume of blood samples for research analyses taken at each sampling point would not exceed 40 ml.

#### 12 STATISTICS

#### 12.1 Number of Participants
The OxAMI-PICSO study aims to investigate the potential benefit of PICSO in a highly selected population

of STEMI patients. In line with the data reported by Sayeed et al in a previous metanalysis on 7 studies

about PICSO application in animal models, the recently published Prepare-RAMSES study also observed a

30% reduction in IS in the treatment arm, however such reduction was not statistically significant in

comparison to the control arm [19]. The study, however could still show a benefit of PICSO in terms of IS

reduction at six months follow up in the subgroup of patients receiving high PICSO quantity. The study,

however, was significantly hampered by the inclusion of relative low risk patients and by a small sample

size. The author managed indeed to deliver full PICSO treatment only in 63% of the initial planned cohort

(12 patients, of the 30 planned, received a prolonged treatment with PICSO) [22].

In order to address the first limitation of the Prepare-RAMSES study, OxAMI-PICSO study will select

patients with a prestenting higher IMR. In this way PICSO is meant to be applied only in a population at

higher risk and highly likely to get benefit from its application.

In this regard assuming that the stricter inclusion criteria may allow to detect a substantial benefit from

PICSO compared to the control group and expecting that this will allow to achieve a significant 29%

reduction in IS as shown in Sayeed's metanalysis [19], we initially calculated a final sample size of 12

patients with complete final data per each group with an interval of confidence at 95% and a 80% power.

However considering that this was the final same sample size enrolled in the Prepare-RAMSES study,

initially meant to recruit 30 patients per arm, we propose to double the actual sample size from 12 to 25

per arm.

Allowing for participants who do not wish to undergo repeat cardiac catheterisation, or cardiac MRI, we

anticipate that approximately 75 patients may be recruited to the study in order to achieve full

participation and complete follow up in 25 subjects.

12.2 Analysis of Endpoints

In keeping with our usual practice we will obtain expert statistical advice from the Centre for Statistics in

Medicine (or equivalent) for each specific task. Summary statistics, including means, medians, and

26 February 2018 Version 5.0

variances, will be calculated at each time point and for each type of data (e.g. parameters derived from

coronary physiology and CMR). The distribution of the levels will be described. It may be necessary to log

transform the data before further statistical analysis. For each parameter an analysis of variance will be

carried out at each time point.

Control group in OxAMI-PICSO study is represented by a highly matched group of patients underwent to

primary PCI, with a prestenting IMR > 40 and with available 24 hours recath and 24-48 hours/6 months

CMR data. Matching will be performed by application of a propensity score matching analysis including

the following predictors in the model: age, sex, pain to wire time, thrombotic burden (assessed as

angiographic thrombus score), thrombus aspiration performance, stent volume, glycoprotein IIbIIIa

inhibitors adoption.

13 DATA MANAGEMENT

13.1 Source Data

Source documents are where data are first recorded, and from which participants' CRF data are obtained.

These include, but are not limited to, hospital records (from which medical history and previous and

concurrent medication may be summarised into the CRF), clinical and office charts, laboratory and

pharmacy records, diaries, microfiches, radiographs, and correspondence.

CRF entries will be considered source data if the CRF is the site of the original recording (e.g. there is no

other written or electronic record of data). All documents will be stored safely in confidential conditions.

On all trial-specific documents, other than the signed consent, the participant will be referred to by the

trial participant number/code, not by name.

13.2 Access to Data

Direct access will be granted to authorised representatives from the Sponsor, host institution and the

regulatory authorities to permit trial-related monitoring, audits and inspections.

Medical Device Clinical Investigation Protocol Template version DRAFT

© Copyright: The University of Oxford and Oxford University Hospitals NHS Trust 2014


13.3 Data Recording and Record Keeping

Study data will be entered on case record forms (CRF). The department SOP on database design will be

followed. Data will be uploaded into SPSS or equivalent statistical software for statistical analysis. The

participants will be identified by a study specific participant number in any database. The name and any

other identifying detail will NOT be included in any study data electronic file. All data will be made non

patient-identifiable as soon as is practical to do so via the participant ID.

14 QUALITY ASSURANCE PROCEDURES

The trial will be conducted in accordance with the current approved protocol, ICH GCP, relevant

regulations and standard operating procedures.

Regular monitoring will be performed by the sponsor according to ICH GCP. Data will be evaluated for

compliance with the protocol and accuracy in relation to source documents. Following written standard

operating procedures, the monitors will verify that the clinical trial is conducted and data are generated,

documented and reported in compliance with the protocol, GCP and the applicable regulatory

requirements.

15 SERIOUS BREACHES

A serious breach is defined as "A breach of GCP or the trial protocol which is likely to affect to a significant

degree -

(a) the safety or physical or mental integrity of the subjects of the trial; or

(b) the scientific value of the trial".

In the event that a serious breach is suspected the Sponsor must be contacted within 1 working day. In

collaboration with the C.I., the serious breach will be reviewed by the Sponsor and, if appropriate, the

Sponsor will report it to the REC committee, Regulatory authority and the NHS host organisation within

seven calendar days.

16 ETHICAL AND REGULATORY CONSIDERATIONS

16.1 Specific Ethical Considerations for participants in emergency situations

Research in emergency situations is ethically complex because of the urgent nature of the interventions

and the often severely compromised capacity of the patient. The processes of enrolment and consent

described above, including verbal consent and assent, the involvement of the Advocate represents our

attempt to develop a thorough, ethically justified process that both protects patients' rights and interests

and enables important research to be done. These processes have been developed in the light of and

guided by the provisions laid out in the Mental Capacity Act with special reference to Section 32(9).

16.2 Possible risks and/or discomfort for patient

Patients referred for cardiac catheterization and PCI will undergo this procedure as would routinely be

performed. Patients will therefore be consented for the standard of care procedure and its associated

risks.

Overall the PCI procedure time may be lengthened by around 20 minutes to complete the selected study

procedures (cardiac physiological measurements + PICSO catheter placement). In the context of a PCI

procedure that typically last approximately 60 minutes; the additional time taken should not result in any

clinically significant difference to the participants. Very occasionally this additional time can result in some

back discomfort for patients having to lie on the angiography bed for the additional time period.

CMR is an established cardiac imaging technique in our institution and is generally very well tolerated.

Specific considerations for safety are reflected by the additional exclusion criteria listed in section 7.3. All

local protocols will be adhered to and only fully trained staff will carry out procedure according to

departmental SOPs.

16.3 Collaboration and Partnership with Commercial Companies

The University of Oxford, the Oxford University Hospitals NHS Trust (OUHT) and the OxAMI-PICSO study

may work in partnership with, and receive support from, commercial companies who provide the devices

and technologies related to PCI and other research investigations. As part of this partnership we may make available research data to the company specifically related to the use of their device or technology. All data will be supplied in a fully anonymised format and participants would not be identifiable from this.

## 16.4 Feasibility

## 16.4.1 Facility

The Oxford Heart Centre is a state-of-the-art facility which incorporated services in cardiology and cardiac surgery. The cardiac catheter laboratories are fully equipped to support these studies.

### 16.5 Declaration of Helsinki

The Investigator will ensure that this trial is conducted in accordance with the principles of the Declaration of Helsinki.

## 16.6 ICH Guidelines for Good Clinical Practice

The Investigator will ensure that this trial is conducted in full conformity with relevant regulations and with the ICH Guidelines for Good Clinical Practice (CPMP/ICH/135/95) July 1996.

## 16.7 Medical Device regulations

The Investigator will ensure that this trial is conducted in full conformity with:

- European Commission Medical Device Guidelines relating to the application of the EU Directives
   on Medical Devices
- Guide to European Medical Device Trials and BS EN ISO 14155

### 16.8 Approvals

26 February 2018 Version 5.0

The protocol, informed consent form, participant information sheet and any proposed advertising material

will be submitted to an appropriate Research Ethics Committee (REC), and host institution(s) for written

approval.

The Investigator will submit and, where necessary, obtain approval from the above parties for all

substantial amendments to the original approved documents.

16.9 Reporting

The CI shall submit once a year throughout the clinical trial, or on request, an Annual Progress Report to

the REC, host organisation and Sponsor. In addition, an End of Trial notification and final report will be

submitted to the REC, host organisation and Sponsor.

16.10 Participant Confidentiality

The trial staff will ensure that the participants' anonymity is maintained. The participants will be identified

only by initials and a participants ID number on the CRF and any electronic database. All documents will

be stored securely and only accessible by trial staff and authorised personnel. The trial will comply with

the Data Protection Act, which requires data to be anonymised as soon as it is practical to do so.

16.11 Potential Benefits

The information derived from coronary pressure/flow measurements is often very useful to the

interventional cardiologist in optimising PCI strategy, and the use of vasodilators (e.g. adenosine) as part

of the coronary pressure/flow measurements often results in useful clinical improvements in coronary

flow.

Finally PICSO treatment, according to pre-clinical literature evidences, is expected to provide a benefit in

terms of infarct size reduction. According to animal models this advantage should amount around a 29%

in reduction of the infarcted area. The application of PICSO treatment in a highly selected, high risk

population of STEMI patients should amplify the potential benefits of this therapy.

Medical Device Clinical Investigation Protocol Template version DRAFT © Copyright: The University of Oxford and Oxford University Hospitals NHS Trust 2014 **CONFIDENTIAL** 

### 17 FINANCE AND INSURANCE

# 17.1 Funding

The study will be supported by British Heart Foundation, NIHR Biomedical Research Centre programme. Miracor Medical Systems will support the study by providing PICSO catheters, PICSO Impulse Console and an unrestricted grant.

#### 17.2 Insurance

NHS bodies are legally liable for the negligent acts and omissions of their employees. If the patient is harmed whilst taking part in a clinical trial as a result of negligence on the part of a member of the study team a liability cover would apply. Non-negligent harm is not covered by the NHS indemnity scheme. The Oxford University Hospitals NHS Trust, therefore, cannot agree in advance to pay compensation in these circumstances. In exceptional circumstances an ex-gratia payment may be offered.

### 18 PUBLICATION POLICY

Data will be owned and supervised by the trust. The Investigators will be involved in reviewing drafts of the manuscripts, abstracts, press releases and any other publications arising from the study. Authors will acknowledge that the study was Funded by British Heart Foundation, NIHR Biomedical Research Centre programme and Miracor Medical Systems. Authorship will be determined in accordance with the ICMJE guidelines and other contributors will be acknowledged. Copies of any publications connected to this study are available on request from the OXAMI-PICSO investigators.

#### 19 REFERENCES

[1] Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, et al. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the

special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI).

Eur Heart J. 2014 Aug 29.

- [2] Roe MT, Ohman EM, Maas AC, Christenson RH, Mahaffey KW, Granger CB, et al. Shifting the openartery hypothesis downstream: the guest for optimal reperfusion. J Am Coll Cardiol. 2001 Jan;37(1):9-18.
- [3] Niccoli G, Burzotta F, Galiuto L, Crea F. Myocardial no-reflow in humans. J Am Coll Cardiol. 2009 Jul 21;54(4):281-92.
- [4] De Maria GL, Patel N, Kassimis G, Banning AP. Spontaneous and procedural plaque embolisation in native coronary arteries: pathophysiology, diagnosis, and prevention. Scientifica (Cairo). 2013; 2013: 36424
- [5] Ng MK, Yong AS, Ho M, Shah MG, Chawantanpipat C, O'Connell R, et al. The index of microcirculatory resistance predicts myocardial infarction related to percutaneous coronary intervention. Circ Cardiovasc Interv. 2012 Aug 1;5(4):515-22.
- [6] Fearon WF, Shah M, Ng M, Brinton T, Wilson A, Tremmel JA, et al. Predictive value of the index of microcirculatory resistance in patients with ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2008 Feb 5;51(5):560-5.
- [7] McGeoch R, Watkins S, Berry C, Steedman T, Davie A, Byrne J, et al. The index of microcirculatory resistance measured acutely predicts the extent and severity of myocardial infarction in patients with ST-segment elevation myocardial infarction. JACC Cardiovasc Interv. 2010; **3**(7): 715-22.
- [8] Fearon WF, Low AF, Yong AS, McGeoch R, Berry C, Shah MG, et al. Prognostic value of the Index of Microcirculatory Resistance measured after primary percutaneous coronary intervention. Circulation. 2013 Jun 18;127(24):2436-41.
- [9] Pratt FH. The nutrition of the heart though the vessels of thebesius and the coronary veins. Am J Physiol. 1898;1:86.

- [10] Lazar HL, Rajaii A, Roberts AJ. Reversal of reperfusion injury after ischemic arrest with pressure-controlled intermittent coronary sinus occlusion. J Thorac Cardiovasc Surg. 1988 Apr;95(4):637-42.
- [11] Lazar HL. Advantages of pressure-controlled intermittent coronary sinus occlusion over left ventriclepowered coronary sinus retroperfusion. Ann Thorac Surg. 2001 Jan;71(1):402.
- [12] Bedi HS, Suri A, Kalkat MS, Sengar BS, Mahajan V, Chawla R, et al. Global myocardial revascularization without cardiopulmonary bypass using innovative techniques for myocardial stabilization and perfusion.

  Ann Thorac Surg. 2000 Jan;69(1):156-64.
- [13] Martin JS, Byrne JG, Ghez OY, Sayeed-Shah U, Grachev SD, Laurence RG, et al. LV-powered coronary sinus retroperfusion reduces infarct size in acutely ischemic pigs. Ann Thorac Surg. 2000 Jan;69(1):84-9.
- [14] Ido A, Hasebe N, Matsuhashi H, Kikuchi K. Coronary sinus occlusion enhances coronary collateral flow and reduces subendocardial ischemia. Am J Physiol Heart Circ Physiol. 2001 Mar;280(3):H1361-7.
- [15] Beatt KJ, Serruys PW, de Feyter P, van den Brand M, Verdouw PD, Hugenholtz PG. Haemodynamic observations during percutaneous transluminal coronary angioplasty in the presence of synchronised diastolic coronary sinus retroperfusion. Br Heart J. 1988 Feb;59(2):159-67.
- [16] Weigel G, Kajgana I, Bergmeister H, Riedl G, Glogar HD, Gyongyosi M, et al. Beck and back: a paradigm change in coronary sinus interventions--pulsatile stretch on intact coronary venous endothelium. J Thorac Cardiovasc Surg. 2007 Jun;133(6):1581-7.
- [17] Mohl W, Mina S, Milasinovic D, Kasahara H, Wei S, Maurer G. Is activation of coronary venous cells the key to cardiac regeneration? Nat Clin Pract Cardiovasc Med. 2008;5:528-30.
- [18] Khattab AA, Stieger S, Kamat PJ, Vandenberghe S, Bongoni A, Stone GW, et al. Effect of pressure-controlled intermittent coronary sinus occlusion (PICSO) on myocardial ischaemia and reperfusion in a closed-chest porcine model. EuroIntervention. 2013 Jul;9(3):398-406.

[19] Syeda B, Schukro C, Heinze G, Modaressi K, Glogar D, Maurer G, et al. The salvage potential of coronary sinus interventions: meta-analysis and pathophysiologic consequences. J Thorac Cardiovasc Surg. 2004 Jun;127(6):1703-12.

[20] Mohl W, Glogar DH, Mayr H, Losert U, Sochor H, Pachinger O, et al. Reduction of infarct size induced by pressure-controlled intermittent coronary sinus occlusion. Am J Cardiol. 1984 Mar 15;53(7):923-8.

[21] Van de Hoef TP, Nolte F, Delewi R, Henriques JP, Spaan JA, Tijssen JG, et al. Intracoronary hemodynamic effects of pressure-controlled intermittent coronary sinus occlusion (PICSO): results from the First-In-Man Prepare PICSO Study. J Interv Cardiol. 2012 Dec;25(6):549-56.

[22] van de Hoef TP, Nijveldt R, van der Ent M, Neunteufl T, Meuwissen M, Khattab A, et al. Pressure-controlled intermittent coronary sinus occlusion (PICSO) in acute ST-segment elevation myocardial infarction: results of the Prepare RAMSES safety and feasibility study. EuroIntervention. 2015; 11: 37-44.

[23]. Cuculi F, Dall'Armellina E, Manlhiot C, De Caterina AR, Colyer S, Ferreira V, et al. Early change in invasive measures of microvascular function can predict myocardial recovery following PCI for ST-elevation myocardial infarction. Eur Heart J. 2014;35:1971-80.

[24] Bonderman D, Teml A, Jakowitsch J, Adlbrecht C, Gyongyosi M, Sperker W, et al. Coronary no-reflow is caused by shedding of active tissue factor from dissected atherosclerotic plaque. Blood. 2002; 99: 2794-800

- [25] Bobryshev YV, Farnsworth AE, Lord RS. Expression of vascular endothelial growth factor in aortocoronary saphenous vein bypass grafts. Cardiovascular surgery (London, England). 2001; 9: 492-8.
- [26] Porter KE, Turner NA. Statins for the prevention of vein graft stenosis: a role for inhibition of matrix metalloproteinase-9. Biochemical Society transactions. 2002; 30: 120-6.

- [27] Wang AY, Bobryshev YV, Cherian SM, Liang H, Tran D, Inder SJ, et al. Expression of apoptosisrelated proteins and structural features of cell death in explanted aortocoronary saphenous vein bypass grafts. Cardiovascular surgery (London, England). 2001; 9: 319-28
- [28] Khachigian LM, Fahmy RG, Zhang G, Bobryshev YV, Kaniaros A. c-Jun regulates vascular smooth muscle cell growth and neointima formation after arterial injury. Inhibition by a novel DNA enzyme targeting c-Jun. The Journal of biological chemistry. 2002; 277: 22985-91.
- [29] Bhindi R, Brieger D, Ishii H, Di Girolamo N, Kumar RK, Khachigian LM, et al. Fibroblast growth factor 2 and the transcription factor Egr-1 localise to endothelial cell microvascular channels in human coronary artery occlusion. Thrombosis and haemostasis. 2005; 93: 172-4.

## 20. APPENDIX A: SCHEDULE OF PROCEDURES IN PICSO GROUP

| Procedures | PICSO group | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | During PCI | | | | 6 | 24 | 48 | 6 |
| | Pre-PCI | Start of procedure | PICSO start | End of PCI | PICSO stop | hours | hours | hours | months |
| Verbal assent | X | | | | | | | | |
| Blood samples | | Х | Х | Х | Х | Х | Х | Х | Х |
| PICSO | | | Х | х | Х | | | | |
| Coronary physiology measurements (IMR, CFR, FFR) | | Х | | Х | | Х | | | |
| Informed written consent | | | | | | Х | | | |
| Coronary angiogram with coronary physiology measurements (IMR, CFR, FFR) | | | | | | | Х | | |
| CMR | | | | | | | | Х | Х |
| ECG | Х | | | Х | | Х | | | |
| Echocardiography | | | | | | | Х | | |
| Medical history Demographic data collection | | | | | | | | Х | |

26 February 2018 Version 5.0

# 21. APPENDIX B: SCHEDULE OF PROCEDURES IN NON-PICSO GROUP

| Procedures | NON-PICSO group | | | | | | |
|---|---|---|---|---|---|---|---|
| | Pre-PCI | Dur | ing PCI | 6 hours | 24 hours | 48 hours | 6 months |
| | | Start of procedure | End of PCI | | | | |
| Verbal assent | Х | | | | | | |
| Blood samples | | Х | Х | Х | Х | Х | Х |
| Coronary physiology measurements (IMR, CFR, FFR) | | Х | Х | | | | |
| Informed written consent | | | | Х | | | |
| ECG | Х | | Х | Х | | | |
| Echocardiography | | | | | Х | | |
| Medical history Demographic data collection | | | | | | Х | |